CLINICAL TRIAL: NCT03826017
Title: A 12 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Catechin High Contain Greentea Extract on Improvement of Cognitive Function
Brief Title: Efficacy and Safety of Catechin High Contain Greentea Extract on Improvement of Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Young Chul Chung, Professor of Psychiatry, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RNO-CF-EG
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Cognitive Function
Keywords: Catechin high contain greentea extract; Cognitive Function

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catechin high contain greentea extract (Experimental): Catechin high contain greentea extract for 260 mg/day 12 weeks.
  Interventions: Dietary Supplement: Catechin high contain greentea extract
- Placebo (Placebo Comparator): Placebo for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Catechin high contain greentea extract — Catechin high contain greentea extract 260 mg/day for 12 weeks.
  Arms: Catechin high contain greentea extract
Dietary Supplement: Placebo — Placebo for 12 weeks.
  Arms: Placebo

SUMMARY:
This study was the efficacy and safety of Catechin high contain greentea extract on improvement of Cognitive Function

DETAILED DESCRIPTION:
This study was a 12 weeks, randomized, double-blind, placebo-controlled human trial to evaluate. 80 subjects were participated in Catechin high contain greentea extract or placebo group. To evaluate the changes of the evaluation items when Catechin high contain greentea extract was taken 12 weeks compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Those who are at least 60 years of age at screening
* Those who have Korean Mini-Mental Status Examination(K-MMSE) result 25-28 points
* Those who agree to voluntary participation and to comply with the Notice after fully hearing and understanding the details of this human trial

Exclusion Criteria:

* Those with a past history of treatment with Axis I disorder in SCID(Structured Clinical Interview for DSM-IV) which is a structured clinical interview in the Diagnostic and Statistical Manual of Mental Disorders at Screening or who have been treated within the last 3 years
* Those with alcohol abuse or dependence within the last 3 months
* Those who have clinically significant following severe illness (Epilepsy, mental retardation, brain nervous system diseases, endocrine diseases, blood / malignant tumors, cardiovascular diseases, Crohn's disease, etc.)
* Those with a history of clinically significant hypersensitivity to green tea
* Those taking medicines, health functional foods or herbal medicines related to improvement of cognitive function and memory within 1 month before screening
* Those who ingested green tea extract's health functional food within 1 month before screening
* Those who whole blood donation within 1 months before the first ingestion or Component blood donation within 2 weeks
* Those who participate in other human tiral within 3 months
* Those who shows the following results in the Laboratory test

  * AST, ALT > 3 times upper limit of normal range
  * Other significant laboratory test opinion
* Those who is deemed unsuitable for participating in the human trial due to other reasons

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Changes of Visual learning test | 12 weeks
  Visual learning test was measured in baseline and 12 week.
Changes of Korean Version of the Montreal Cognitive Assessment(MoCA-K) | 12 weeks
  Korean Version of the Montreal Cognitive Assessment(MoCA-K) was measured in baseline and 12 week. The cognitive function evaluation using the Montreal Cognitive Assessment(MoCA-K) is a total of 8 items, and evaluates cognitive functions such as time / execution power, vocabulary, memory, attention, sentence, abstraction, delayed recall, and orientation.
  Time / execution power's total score is 5 points, vocabulary's total score is 3 points, attention's total score is 3 points, sentence's total score is 3 points, abstraction's total score is 2 points, delayed recall's total score is 5 points, orientation's total score is 6 points. It takes about 10 minutes to complete, and the total score is 30 points and total score make sum score. A score of 23 points or more is regarded as normal. If you have less than 6 years of education, add 1 point.

SECONDARY OUTCOMES:
Changes of Auditory continuous performance test | 12 weeks
  Auditory continuous performance test was measured in baseline and 12 week.
Changes of Verbal learning test | 12 weeks
  Verbal learning test was measured in baseline and 12 week.
Changes of Visual working memory test | 12 weeks
  Visual working memory test was measured in baseline and 12 week.
Changes of Perceived stress scale(PSS) | 12 weeks
  Perceived stress scale(PSS) was measured in baseline and 12 week. It consists of 10 questions. Each question is evaluated from 0 (none) to 4 (very often), and 4 items (4, 5, 7, 8) are scored back and added to the remaining questions. The duration of the last month should be presented before implementation (if the duration is longer, the predictability is lowered).
Changes of Beck Depression Inventory(BDI) | 12 weeks
  Beck Depression Inventory(BDI) was measured in baseline and 12 week. It consists of 21 items including cognitive, emotional, synchronous, and physical symptoms of depression. The total score ranges from 0~63 points for each question. Beck Depression Inventory(BDI) score is 0 ~ 9 points non-depression, 10 ~ 15 is mild depression, 16 ~ 23 is moderate depression, and 24 ~ 63 is severe depression.
Changes of Brain-derived neurotrophic factor(BDNF) | 12 weeks
  Brain-derived neurotrophic factor(BDNF)(pg/mL) was measured in baseline and 12 week.
Changes of Total antioxidant status(TAS) | 12 weeks
  Total antioxidant status(TAS) was measured in baseline and 12 week.

CONTACTS AND LOCATIONS:
Overall Officials: Young-chul Chung, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Department of Psychiatry, Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea